CLINICAL TRIAL: NCT01915329
Title: Effects of Repetitive Electric Sensory Stimulation on Sensorimotor Performance and Pain Intensity in Complex Regional Pain Syndrome Type I
Brief Title: Effects of Repetitive Electric Sensory Stimulation (RSS) as Intervention in Complex-regional-pain-syndrome Type I (CRPS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr. med Christoph Maier, Head Dep. of Pain Medicine, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RSS_2012
Record Dates: First submitted 2013-05-13; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Complex Regional Pain Syndrome Type I of the Upper Limb
Keywords: CRPS; repetitive sensory stimulation; cortical reorganization; 2-point-discrimination
MeSH Terms: conditions — Reflex Sympathetic Dystrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum-RSS (Experimental): RSS Stimulation with high frequency electric pulses
  Interventions: Device: RSS (repetitive sensory stimulation)
- Sham-RSS (Sham Comparator): Sham RSS Stimulation (no pulses are transmitted)
  Interventions: Device: SHAM-RSS

INTERVENTIONS:
Device: RSS (repetitive sensory stimulation) — RSS is a high frequency electrical stimulation protocol delivered to the peripheral nerves (median and ulnar nerve) of the hand. The signals are generated by a TENS-stimulator and are conveyed to each finger of the hand via a custom-made hand-shaped device with conductive contacts at each fingertip and at the palmar base.
  In case of the sham-stimulation no pulses are transmitted.
  Arms: Verum-RSS
Device: SHAM-RSS — The same device as in the RSS intervention is used, but no electrical stimuli are transmitted.
  Arms: Sham-RSS

SUMMARY:
The purpose of this study is to test a specific nerve stimulation protocol as therapeutic option in patients diagnosed with CRPS (complex regional pain syndrome) of the upper extremity.

DETAILED DESCRIPTION:
A specific high frequency electric stimulation is conveyed at 5 days to the affected hand. Each stimulation session lasts 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CRPS Type I

Exclusion Criteria:

* intolerable hyperalgesia
* lesions at the fingertips
* high grade digit contracture
* central neurologic disorders
* psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
static tactile 2-point-discrimination threshold | before and after the 5 day stimulation phase with a minimum time of 1h between measurements and start/end of the stimulation (day1 pre and day 5 post)
  Thresholds on the tip of the index finger of both hands are assessed using the method of constant stimuli. One single needle and seven pairs of needles with different spacings are tested in randomized order. After each presentation, the subject has to report the sensation of one or two needles by answering immediately "one" or "two." Each distance is presented eight times resulting in 64 single decisions. The summed responses are plotted against distance as a psychometric function for absolute threshold and get fitted by a binary logistic regression. Threshold are taken from the fit at the distance at which 50% correct answers are given.

SECONDARY OUTCOMES:
pain intensity | before and after the 5 day stimulation phase with a minimum time of 1h between measurements and start/end of the stimulation (day1 pre and day 5 post)
  Pain intensity is rated by the patient on a 11-point numerical rating scale (NRS). Pain intensity is rated before the start of the 5 day stimulation phase (baseline,pre) and at the end (post, in combination with the other outcome measures). Additionally pain intensity is rated directly before the start of each daily stimulation session and immediately after each session of 45 minute duration.

OTHER OUTCOMES:
somatosensory evoked potentials | before and after the 5 day stimulation phase with a minimum time of 1h between measurements and start/end of the stimulation (day1 pre and day 5 post)
  Somatosensory evoked potentials after electrical paired pulse median nerve stimulation are recorded. The median nerve is stimulated by innocuous paired electrical pulses conveyed to the nerve by a block electrode placed on the wrist. For correct positioning the subject has to report a prickling sensation in thumb, index and middle finger. Stimulation intensity is choosen to induce a small muscular twich at the thenar muscles. SEP recordings are done with a 3-electrode array. Two electrodes are fixed on the scalp over the left and right somatosensory cortex. The third (reference) electrode is fixed over the midfront. SEP signals get amplified and filtered and digitized in a PC.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pain Medicine, BG Universitätsklinikum Bergmannsheil GmbH, Bochum, North Rhine-Westphalia, Germany